CLINICAL TRIAL: NCT06263387
Title: Results From a Nationwide Cohort Temporary Utilization Authorization (ATU) of First-line Acute Myeloid Leukemia (AML) Patients Ineligible for Intensive Chemotherapy (IC),Treated in France With Venetoclax Azacitidine
Brief Title: Results From a French Temporary Utilization Authorization of First-line Acute Myeloid Leukemia (AML) Patients Ineligible for Intensive Chemotherapy (IC), Treated With Venetoclax Azacitidine
Acronym: VENAZA
Status: Recruiting | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Acute Leukemia French Association (Other)
Responsible Party: Sponsor
Other Study IDs: FILObsLAM_VENAZA
Record Dates: First submitted 2023-12-14; First posted 2024-02-16 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Following the results of the phase 1b and the phase 3 studies, Venetoclax/Azacitidine (VEN/AZA) was available in France for newly diagnosed AML patients ineligible-IC patients through the early access program the so-called ATU program.

Venetoclax (VEN) has been available in France through the ATU since Feb 2021 and through the current post-ATU schema from the point of marketing authorization approval and up to the pending publication of reimbursement and price. Between February 15, 2021, and June 30, 2021, 285 requests for ATU were made to the pharmaceutical company (Abbvie) and led to the initiation of treatment of more than 230 patients. At the end of ATU period, all these 230 ATU patients continued to be treated by VEN/AZA as part of the current post-ATU period. Healthcare professionals and health care decision makers need real world data to better understand the benefit/risk profile of treatment. Early access to treatment in France is close to real-life setting condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* treatment with VEN-AZA for newly diagnosed AML and ineligible to intensive chemotherapy
* Treatment in the named-patients program (ATU)

Exclusion Criteria:

* Treatment with VEN-AZA for previously treated AML

  * Prior treatment for preexisting hematological malignancies other that AML, including AZA is not an exclusion criteria
  * HYDROXYCARBAMIDE given for AML is not an exclusion criteria
  * AZA started before VEN for AML is not an exclusion criteria
* Opposition to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients with de novo AML, ineligible for intensive chemotherapy, which received VENAZA in the ATU program between 02/15/2021 and 06/30/2021
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
characterize the overall response rate, in patients treated by Venetoclax/Azacitidine (VEN/AZA), in real life cohort | 18 months (since Cycle 1 Day 1)
  1. Rate of complete remission and complete remission with incomplete hematologic recovery (CR/CRi),
  2. Rate of morphological leukemia free state (MLFS)
  3. Rate of CR/CRi rate with negative minimal residual disease (MRD) assessed by flow cytometry (FCT) and/or molecular techniques if available
characterize the overal survival (OS) in patients treated by Venetoclax/Azacitidine (VEN/AZA), in real life cohort | 18 months (since Cycle 1 Day 1)
  rate of OS according to the 2022 European LeukemiaNet (ELN)
characterize the event free survival (EFS) in patients treated by Venetoclax/Azacitidine (VEN/AZA), in real life cohort | 18 months (since Cycle 1 Day 1)
  rate of EFS according to the 2022 European LeukemiaNet (ELN)

SECONDARY OUTCOMES:
characterize the incidence and relatedness of serious adverse events (SAE), in patients treated by Venetoclax/Azacitidine (VEN/AZA), in real life | 18 months (since Cycle 1 Day 1)
  description of grade 3/4 SAE and death according to CTCAE v5.
describe the management of Venetoclax/Azacitidine (VEN/AZA) in a real -life cohort of patient. | 18 months (since Cycle 1 Day 1)
  daily dose and duration of Venetoclax and Azacitidine description of Venetoclax and Azacitidine dose modification description of Venetoclax and Azacitidine duration

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain GARCIAZ, MD-PhD, Principal Investigator — French Innovative Leukemia Organisation
Locations (42):
- France (42):
  - Amiens CHU, Amiens
  - Angers CHU, Angers
  - Avignon CH, Avignon
  - Bayonne CH, Bayonne
  - Besançon CHU, Besançon
  - Brest CHU, Brest
  - Caen CHU, Caen
  - CERGY PONTOISE - CH René Dubos, Cergy-Pontoise
  - Hôpital d'Instruction des Armées PERCY, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Corbeil-Essonnes - Ch Sud Francilien, Corbeil-Essonnes
  - Créteil CHU HENRI MONDOR, Créteil
  - Dijon CHU, Dijon
  - Grenoble CHU, Grenoble
  - Le Mans CH, Le Mans
  - CHU Lille, Lille
  - Limoges CHU, Limoges
  - Lyon sud CHU, Lyon
  - Marseille IPC, Marseille
  - Meaux CH de l'Est francilien, Meaux
  - METZ-THIONVILLE CHR- Hôpital de Mercy, Metz
  - Montpellier - Chu Saint Eloi, Montpellier
  - Nantes CHU, Nantes
  - Nice CHU, Nice
  - Nimes CHU, Nîmes
  - Paris La Pitié salpetrière, Paris
  - Paris Necker, Paris
  - Paris Saint Louis, Paris
  - Bordeaux CHU, Pessac
  - Reims CHU, Reims
  - Rennes CHU, Rennes
  - roubaix CH, Roubaix
  - Centre de Lutte Contre le Cancer H. Becquerel, Rouen
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Saint Quentin CH, Saint-Quentin
  - ICANS - Institut de cancérologie de strasbourg europe, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - Tours CHU, Tours
  - Troyes CH, Troyes
  - Nancy CHU, Vandœuvre-lès-Nancy
  - Versailles CH, Versailles
  - Villejuif IGR, Villejuif

IPD SHARING:
Plan to Share IPD: No